## Arcos® Revision Stem: Evaluation of Clinical Performance

A Retrospective and Prospective Multi-Center Two-Armed Non-Comparative Clinical Investigation on 200 subjects

PROTOCOL Number (Study ID): GBMET.CR.US19.12
PROTOCOL data and version: March 18, 2015, Version. 6
NCT Number: 01820611

Arcos Study

## **1 STUDY SYNOPSIS**

| TITLE | Arcos Revision Stem: Evaluation of Clinical Performance |
|---|---|
| CIP ID | GBMET.CR.US19 |
| SPONSOR | Original: Biomet Administratively transferred: Zimmer GmbH, Zählerweg 4, 6300 Zug, Switzerland |
| MANUFACTURER | Biomet Orthopedics |
| STUDY DEVICE (S) | Arcos Modular Revision Femoral System |
| | The primary purpose of this study is to evaluate the clinical performance of the Arcos Revision Stem system, determine the stability of the implants, and evaluate any relationship between bone defect level and the success of the Arcos Stem. |
| | Primary Endpoints: |
| OBJECTIVE/ENDPOINTS | - Survivorship and revision rate up to 5 years |
| | Secondary Endpoints: |
| | <ul> <li>Stability and Fixation of Arcos Hip by radiographic assessment, Relationship between bone defect level, Oxford hip score and Harris hip score postoperative</li> <li>Adverse events, complications</li> </ul> |
| POPULATION | 200 Patients: 100 with BoneMaster HA, 100 without BoneMaster HA Up to ten sites will be used to fulfill enrollment to this study All cases enrolled will be those implanted with either the Cone, Broached, or Calcar Proximal Body and one of the five distal options (Slotted, Bullet-tip, Interlocking, STS, or ETO). |
| ELIGIBILITY | To be included in the study, a patient have received a revision total hip arthroplasty with the Arcos system. The Arcos system is to be used in accordance to the indications for use and contraindications detailed in the approved labeling of the device. |
| | Inclusion Criteria |
| INCLUSION/EXCLUSION<br>CRITERIA | Patients will be included in this study if they received the Arcos Modular Femoral Revision System per the approved indications for use for Arcos specifically. - Patients undergoing Revision of previously failed |
| | total hip arthroplasty. |

Arcos Study

| | The Arcos™ Modular Femoral Revision System hip components are single-use implants, intended for uncemented use only. Only subjects who have received the Arcos Revision Stem System will be included in this outcomes study. Exclusion Criteria Absolute contraindications include: active infection, sepsis, and osteomyelitis. Relative contraindications include: - Uncooperative patient or patient with neurologic disorders who are incapable of following directions - Osteoporosis - Metabolic disorders which may impair bone formation - Osteomalacia - Distant foci of infections which may spread to the implant site - Rapid joint destruction, marked bone loss or bone |
|---|---|
| | resorption apparent on roentgenogram - Vascular insufficiency, muscular atrophy, or neuromuscular disease. |
| | Additionally, all vulnerable subjects (minors, limited or non-readers; adult subjects who cannot consent for themselves; and, pregnant women) will be excluded from participation in this study. |
| STUDY DESIGN | Retrospective and Prospective Multi-Center Two Armed Non-Comparative Trial |
| CLINICAL PHASE | Post-Market |
| NUMBER OF SUBJECTS | 200 Patients - 100 with BoneMaster HA - 100 without BoneMaster HA |
| LENGTH OF STUDY | 5 years (24 months enrolment and 5 years follow up) |
| MATERIAL AND<br>METHODS | Case Report Forms will be completed at 6-12 months, 2-3 years and 5 years post-operatively. |

## **2 STATISTICAL ANALYSIS PLAN**

Arcos Study

**DATA REPORTING** 

The sponsor will present an annual report to the investigators that will include a summary of the

clinical data. The report will contain the results of the Harris Hip at each time point. Also, patient

follow-up will be analyzed throughout the data collection according to the following definition

and equations:

Lost To Follow-Up: 1. Death

2. Revision

3. Consent Rescinded

Percentage Follow-up = # Patients with Follow-Up\_\_\_\_\_ x 100

(Theoretically due – Lost To Follow-Up)

Percentage Accounted for = (# with Follow-Up + Lost To Follow-Up) x 100

Theoretically due

At the end of the data collection, a final report will be compiled that will summarize all data

collected throughout the data collection, complications throughout the course of the data

collection, and general findings.

SAMPLE SIZE JUSTIFICATION

Observational study with 200 Arcos modular femoral revision cases (100 with Bonemaster and

100 without Bonemaster) to assess survivorship and revision rate up to 5 years.

The sample size for this study is based on anticipated sales (1000 during the first year of

commercialization) and expected lost-to-follow-up over the first 5 years, with the goal of having

a reasonable number of cases for evaluating device survival over the first 5 years of follow up.

An article by Frederick Dorey, et.al. (Journal of Arthroplasty, 1(1):63-69, 1986) recommends

having greater than 20 subjects in follow-up when estimating survivorship. Lost to follow-up for

this study is estimated to be 10% per year. Thus, if 100 patients of the Arcos with Bonemaster HA

and 100 cases of Arcos without Bonemaster are enrolled, there will be 59 patients at 5 years of

follow-up for each variant.

Start with 100 cases and assume a loss of 10% per year

o 1 year: 100-10 = 90

Arcos Study

o 2 year: 90-9= 81

o 3 year: 81-8=73

o 4 year: 73-7= 66

o 5 year: 66-7 = 59

59 cases is a reasonable number for evaluating survivorship at 5 years per Dorey, et. al.

Arcos Study